CLINICAL TRIAL: NCT01383044
Title: Banding Ligation With Carvedilol vs. Carvedilol for the Prevention of First Bleeding in Cirrhotics With Moderate Varices
Brief Title: Banding Ligation With Carvedilol Versus Carvedilol for the Prevention of First Bleeding
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: E-DA Hospital (Other)
Responsible Party: IRB, E-DA Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Carvedilol
Record Dates: First submitted 2011-06-16; First posted 2011-06-28 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Variceal Bleeding
Keywords: Carvedilol; Banding ligation with Carvedilol; the efficacy & safety of combining EVL and carvedilol in prevention of first variceal bleeding
MeSH Terms: interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EVL + carvedilol (Experimental): EVL is performed for 2-3 times carvedilol 6.25mg-12.5 mg per day
  Interventions: Procedure: EVL + carvedilol
- carvedilol (Active Comparator): carvedilol 6.25-12.5 mg per day
  Interventions: Drug: carvedilol

INTERVENTIONS:
Procedure: EVL + carvedilol — EVL is performed for 2-3 times carvedilol 6.25mg-12.5 mg per day
  Arms: EVL + carvedilol
Drug: carvedilol — carvedilol 6.25mg-12.5 mg per day
  Arms: carvedilol

SUMMARY:
Endoscopic variceal ligation (EVL) and carvedilol have been documented to be effective in prophylaxis of the first bleeding. The efficacy & safety of combining EVL and carvedilol in prophylaxis of the first bleeding is still unknown. This study aims to investigate the value of combination therapy.

DETAILED DESCRIPTION:
Combination of EVL and β-blocker has been proven effective in the prevention of variceal rebleeding . However, Our previous study showed that combination of EVL and nadolol do not have enhanced effect in the prophylaxis of 1st variceal bleeding as compared with nadolol alone . One of the drawbacks of EVL is esophageal ulcer. On the other hand ,carvedilol, an anti-α beta-blocker, has been proven to be more effective than propranolol in the reduction of portal pressure. Carvedilol has been proven to be more effective than EVL in the prevention of 1st variceal bleeding. The investigators thus conduct a multicenter trial to evaluate whether combination of EVL and carvedilol could be more effective than carvedilol alone in the prophylaxis of 1st esophageal variceal bleeding . The goal of patients receiving EVL is to reduce variceal size, not variceal obliteration, in anticipation for fewer sessions required for each patient and fewer possibility of esophageal ulcer bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhosis with esophageal varices are larger than F2.
2. No history of variceal bleeding.
3. In three months have not implemented preventive esophageal variceal ligation. (4)age 20yrs～75yrs.

Exclusion Criteria:

1. Association with HCC or other cancers .
2. Refractory ascites.
3. Jaundice, bilirubin > 5mg/dl.
4. Encephalopathy.
5. Cr.>3mg/dL.
6. A-V,block bradycardia (PR < 60/mim).
7. Hypotension systolic blood pressure<95/mmHg .
8. Refusal to participate.
9. Carvedilol allergy
10. Second degree-third degree Atrio-ventricular block.
11. Bradycardia.
12. WPWsyndrome
13. Hypotension
14. Psychogenic shock.
15. Asthma. All the patients are randomized based on a random number.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-07-08 (Actual); Primary Completion 2015-07-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
patients with first bleeding | 3 years
  the difference of bleeding episode in both groups.

SECONDARY OUTCOMES:
patients with complications and mortality rates | 3 years
  the difference of complications & survival curve between both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- E-DA hospital, Kaogsiung, Taiwan